CLINICAL TRIAL: NCT05954377
Title: Prospective, Single-center, Randomized, Open Label Study Assessing the Contribution of Telemedicine Monitoring in Addition to Standard Follow-up, Strengthening an Obesity Program in Berry (FRANCE)
Brief Title: Study Assessing the Contribution of Telemedicine Monitoring in Addition to Standard Follow-up of an Obesity Program
Acronym: STROBERRY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STROBERRY
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Obesity
Keywords: obesity; public health; telemedicine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The study concerns patients who ended the 6 months obesity treatment program proposed by the center. At the end of this 6 months care phase, patients will be randomized in 2 groups (ratio 1:1).
  The intervention will be and addition of telemedicine quarterly follow up (remote motivational interviews) to the standard multidisciplinary follow-up post care management program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard multidisciplinary follow-up reinforced with telemedicine (Experimental): Standard annual multidisciplinary follow-up, reinforced with telemedicine (remote quarterly motivational interviews)
  Interventions: Other: Quarterly remote motivational interviews
- Standard multidisciplinary follow up (No Intervention): Standard annual multidisciplinary follow-up without telemedicine follow up

INTERVENTIONS:
Other: Quarterly remote motivational interviews — Remote motivational interview will be in the form of quarterly telephone call (at 3, 6 and 9 months after the start of annual follow up; the patient is seen again at 12 months as part of the annual follow-up) and this for 4 years. It will be performed by medical staff trained in motivational interviewing and who have completed at least 40 hours training in therapeutic education
  Arms: Standard multidisciplinary follow-up reinforced with telemedicine

SUMMARY:
STROBERRY Study is a Prospective, monocentric, randomized, open-label study assessing the contribution of telemedicine, in addition to standard follow-up, strengthening an Obesity program in Berry (France). The principal objective is to study the effectiveness of a follow-up reinforced with telemedicine in addition to the standard multidisciplinary annual follow-up on the rate of patients lost to follow-up after initial or second line management in a multidisciplinary bariatric medical program

DETAILED DESCRIPTION:
Obesity became a major public health issue in France. In 2019, obesity represented 5% of annual costs in health and was responsible of a 2.7% lost in France's Gross Domestic Product. In the scop of french health ministry's recommendations for obese patients'care and the territorial healthcare program; Saint-François' hospital set up 3 healthcare programs: "medical obesity"," interventional" and "post surgery". A very few number of studies aim to asse the efficacity of a long-term telemedicine follow-up after a bariatric medical care program. STROBERRY Study is a Prospective, monocentric, randomized, open-label study assessing the contribution of a long term, telemedical, personalized, educative quarterly, follow-up (4 years follow up), in addition to standard follow-up, strengthening an Obesity program in Berry (FRANCE). The principal objective is to study the effectiveness of a follow-up reinforced with telemedicine in addition to the standard multidisciplinary annual follow-up on the rate of patients lost to follow-up after initial or second line management in a multidisciplinary bariatric medical program

ELIGIBILITY:
Inclusion Criteria:

* Woman or Male aged from 18 to 60 years old included
* Patient in obesity (BMI> or = 30)
* Patient who has completed a multidisciplinary medical program for obesity management, as a first- or second-line intention (after initial obesity management) at the investigating center
* Affiliation to a social security scheme
* Patient informed of the study and who had signed the informed consent form

Non Inclusion Criteria:

* Management of obesity within the framework of an exclusively interventional program, without redirection to a medical program
* Managing obesity as part of a post-operative program
* Pregnant or breastfeeding women
* Patients deprived of liberty
* Patients under legal protection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Rates of patients lost to follow up | 4 years
  Rates of patients lost to follow up measured in both arms and compared 4 years after randomization

SECONDARY OUTCOMES:
The evolution of quality of life, self-esteem and perceived health compared to baseline | 1,2,3 and 4 years
  The evolution of quality of life, self-esteem and perceived health will be measured using the Duke questionnaire, and will be assessed at standard annual visits at 1, 2, 3 and 4 years after randomization
Rate of patients lost to follow-up will be assessed at standard annual visits at 1, 2 and 3 years after randomization | 1,2 and 3 years
  Rate of patients lost to follow-up will be assessed at standard annual visits at 1, 2 and 3 years after randomization
Change in waist circumference (cm) compared with the baseline measurement will be assessed at standard annual visits at 1, 2, 3 and 4 years after randomization. | 1,2,3 and 4 years
  Change in waist circumference (cm) compared with the baseline measurement will be assessed at standard annual visits at 1, 2, 3 and 4 years after randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint-François, Châteauroux, France